CLINICAL TRIAL: NCT02053636
Title: An Open, 3-cohort, Phase II Trial Testing Oral Administration of Lucitanib in Patients With FGFR1-amplified or Non-amplified Estrogen Receptor Positive Metastatic Breast Cancer
Brief Title: A Phase II Trial Testing Oral Administration of Lucitanib in Patients With Fibroblast Growth Factor Receptor (FGFR)1-amplified or Non-amplified Estrogen Receptor Positive Metastatic Breast Cancer
Acronym: FINESSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: Breast International Group (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2-80881-001; 2013-000288-10 (EudraCT Number); BIG 2-13 (Other: BIG)
Record Dates: First submitted 2014-01-24; First posted 2014-02-04 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — E-3810

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lucitanib (Experimental): Hard gelatine capsules of 2,5, 5 and 10 mg or film coated tablets of 5 and 7,5 mg.
  5 to 10 mg orally on a daily basis until unacceptable toxicity according to the investigator, disease progression or withdrawal of consent
  Interventions: Drug: lucitanib

INTERVENTIONS:
Drug: lucitanib

SUMMARY:
The aim of the study is to evaluate the objective response rate (ORR) of single agent lucitanib in metastatic breast cancer patients with FGFR1-amplified, FGFR1-non amplified with 11q amplification, or FGFR1-non amplified without 11q amplification.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast adenocarcinoma.
* Presence of an accessible metastatic lesion for biopsy or at least one archived metastatic tumour sample.
* Prior first-line systemic therapy in the metastatic setting.
* Demonstrated progression of disease by radiological or clinical assessment.
* Female patient, aged ≥18 years old.
* Estimated life expectancy >3 months.
* Normal Left ventricular function
* Adequate haematological, hepatic and renal functions.
* For women with childbearing potential, a negative pregnancy test prior to initiation of the study drug and willingness to use an effective contraception.
* Ability to swallow oral capsules or tablets.

Exclusion Criteria:

* More than two lines of chemotherapy with or without targeted therapy in the metastatic setting.
* Previous treatment with bevacizumab within 3 months of first dose of Investigational Medicinal Product.
* Active central nervous system metastases, cerebral oedema, and/or progressive growth.
* Patients with impaired cardiac function.
* Uncontrolled arterial hypertension
* Patients with history of thrombotic disorders or hereditary risk factors of thromboembolic events
* Serum potassium level below Lower Limit of Normal
* Uncontrolled hypothyroidism.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Every 8 weeks
  Tumor evaluation every 8 weeks throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice André, MD, Study Chair — Institut Gustave Roussy, France; Javier Cortes, MD, Study Chair — Hospital Universitario Vall d'Hebrón, Spain
Locations (29):
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne
  - Westmead Hospital, Westmead
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires St. Luc Oncology - Breast Clinic, Brussels
  - Grand Hôpital de Charleroi Oncologie-Hématologie, Charleroi
  - UZ Leuven Campus Gasthuisberg Dept. of General Medical, Leuven
  - Clinique Sainte-Elisabeth Médecine Interne - Oncologie, Namur
- Canada (3):
  - McGill University Department of Oncologie - Clinical Reserach Program, Montreal
  - Princess Margaret Cancer Centre, Toronto
  - University Health Network - Princess Margaret Hospital, Toronto
- France (3):
  - Institut Claudius Regaud Dpt d'Oncologie Médicale, Toulouse
  - Institut Gustave Roussy Dépt d'oncologie - Cancer du sein, Villejuif
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Kliniken Essen-Mitte Klinik für Senologie - Brustzentrum, Essen
  - KLINIKUM OFFENBACH Klinik für Gynäkologie und Geburtshilfe, Offenbach
  - Klinikum Offenbach, Offenbach
- Hungary (2):
  - Orszagos Onkologiai Intezet Kemoterapia B es Klin.Farm.Oszt., Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum Onkologiai Intezet, Debrecen
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - Istituto Europeo di Oncologia Divisione Sviluppo Nuovi Farmaci per Terapie Innovative, Milan
- Spain (5):
  - H. Valle de Hebrón Servicio de Oncología, Barcelona
  - Hospital Universitario Val d'Hebròn, Madrid
  - MD Anderson Cancer Center Unidad de Investigación Clínica, Madrid
  - H. Ramón y Cajal Servicio de Oncología Médica, Madrid
  - H. Clínico de Valencia Servicio de Hematología y oncología Médica, Valencia
- United Kingdom (4):
  - Western General Hospital Edinburgh Cancer Centre, Edinburgh
  - Royal Marsden Hospital, London
  - The Royal Marsden NHS Trust Dpt of Medicine-Oncology, London
  - Nottingham University Hospitals NHS Trust Department of Clinical Oncology, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Hui R, Pearson RM, Cortes Castan J, Campbell C, Poirot C, Azim HA Jr, Fumagalli R, Lambertini M, Daly F, Arahmani A, Garcia-Perez J, Aftimos PG, Bedard P, Xuereb RG, Loibl S, Loi U, Pierrat MJ, Turner NC, Andre F, Curigliano G. Ann Oncol. 2018 Oct;29(Supplement 8):VIII93. doi: https://doi.org/10.1093/annonc/mdy272.281
- [Background] Liao M, Zhou J, Wride K, Lepley D, Cameron T, Sale M, Xiao J. Population Pharmacokinetic Modeling of Lucitanib in Patients with Advanced Cancer. Eur J Drug Metab Pharmacokinet. 2022 Sep;47(5):711-723. doi: 10.1007/s13318-022-00773-w. Epub 2022 Jul 18. PMID 35844029